CLINICAL TRIAL: NCT06818253
Title: Effects of Glycerol Hyperhydration on Running Economy in Long-Distance Runners
Brief Title: Effect of Glycerol Hyperhydration on Running Economy of Long-distance Runners
Acronym: GHLDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iberoamerican Institute of Sports Science and Human Movement (Other)
Collaborators: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Cesar Octavio Ramos Garcia, PhD, Chief Research Officer (CRO), Iberoamerican Institute of Sports Science and Human Movement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IICDEM-ID-001-2022
Record Dates: First submitted 2025-01-25; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Running; Physical Conditioning, Human
Keywords: Glycerol; athletic performance; sports nutritional sciences; thermoregulation; running
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm glycerol supplementation (Experimental): This arm participated in a crossover design allowed minimizing interindividual variability by using each participant as their own control, evaluating the conditions of (1) hyperhydration with glycerol and (2) water restriction. The main variables evaluated were maximal oxygen consumption (VO₂max), running economy (CE), calculated using the oxygen cost unit (OCU) and caloric cost unit (CCU), as well as body temperature, perception of exertion and sweating rate.
  Interventions: Dietary Supplement: The Effect of Glycerol Supplements

INTERVENTIONS:
Dietary Supplement: The Effect of Glycerol Supplements — The main factor that distinguishes this intervention is first of all the dosage of the dietary supplement and the effects on the variables to be analyzed related to physical performance.

SUMMARY:
The aim of this study was to evaluate the effects of hyperhydration with glycerol on running economy (RE) in trained runners. The main questions sought to be answered are:

1. Does hyperhydration with glycerol improve running economy?
2. Are there beneficial effects on physical performance?

The researchers will conduct a clinical trial with 30 runners (15 men, 15 women) in three sessions. In the first session, VO2peak was determined and running speeds were established for sessions 2 and 3. In the second session, participants performed a stress test. In the second session, participants performed a running test in the euhydrated state under fluid restriction, and in the third session, with glycerol supplementation (22 ml/kg sports drink + 1.2 g/kg glycerol). Variables such as caloric cost unit (CCU), oxygen cost unit (OCU), heart rate (HR), body temperature (BT) and perceived exertion (RPE) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Competitive runners with a minimum record of 4.2 min/km.
2. Age between 18 and 35 years old
3. Apparently healthy athletes
4. Signature of informed consent form

Exclusion Criteria:

1. Presence of comorbidities that could alter the study variables (such as arterial hypertension, hyperthyroidism or heart disease).
2. Consumption of medications or stimulants (such as caffeine or diuretics) 48 hours before the tests.
3. Pregnancy.

   -

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO₂peak) (ml/kg/min) | In the first evaluation session to be held in the first week of a total of 3 weeks of study duration
  Session 1: VO2peak measurements through an incremental treadmill test with 2 km/h speed increments every 3 minutes, maintaining a constant 1% incline. The test started at 6 km/h for all participants and continued until volitional exhaustion
Running economy (CE) | In the first evaluation session to be held in the first week of a total of 3 weeks of study duration
  Test under Hydration Restriction (No-GLY): As a mandatory requirement, participants reported to the laboratory in a euhydrated state (USG: 1.018-1.024) prior to the start of the test, following the criteria outlined in previous research [31]. They ran for 15 minutes on a treadmill at a speed equivalent to 65%-70% of their VO2peak from the first session. During the test, running economy variables such as the caloric cost unit (CCU), oxygen cost unit (OCU), body temperature (BT), rating of perceived exertion (RPE) via the Borg scale, and hydration status were measured.
  Running Economy Calculation:
  i) The caloric cost unit (CCU) was calculated via the following equation [25]: CCU =((VO2 x δ x 1000)/(V x MC)) x 100 where VO2 is the oxygen consumption rate (L/min); δ is the kcal/L of oxygen based on the respiratory exchange ratio (RER); V is the speed (m/min); and MC is the body mass (kg).

SECONDARY OUTCOMES:
Body temperature | Body temperature was measured during sessions 2 (No Gly) and 3 (Gly) at the following times: at minute 0 (prior to the start of each test) and at minutes 5, 10 and 15 during a treadmill test.
  The temperature will be measured during the running economy evaluation with an infrared thermometer (Berrcom® JXB-178).
Perception of exertion | It was applied during the evaluation of the stress tests to determine the Vo2peak and Running Economy.
  The Borg effort perception scale, with a range of scores from 6 to 20, was used during the three sessions, recording the perception of effort in each minute of the test according to the following classification:
  * 6-7: Very very very light
  * 8-9: Very light
  * 10-11: Light
  * 12-13: Regular
  * 14-15: Heavy
  * 16-17: Very heavy
  * 18-19-20: Very very heavy
Sweating rate. | In sessions 1 and 2, urine specific gravity (USG) was assessed, which was one of the key criteria for determining whether subjects could continue in the study without being eliminated.
  Fluctuations in body mass between the different sessions were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Guadalajara, Centro Universitario de Tonalá, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jolicoeur Desroches A, Naulleau C, Deshayes TA, Parent-Roberge H, Pancrate T, Goulet EDB. Effect of Glycerol-Induced Hyperhydration on a 5-kilometer Running Time-Trial Performance in the Heat in Recreationally Active Individuals. Nutrients. 2023 Jan 24;15(3):599. doi: 10.3390/nu15030599. PMID 36771308
- [Derived] Herrera-Amante CA, Garcia-Zepeda G, Garcia-Zepeda CE, Yanez-Sepulveda R, Clemente-Suarez VJ, Lopez-Gil JF, Octavio Ramos-Garcia C. Effects of glycerol hyperhidration on the running economy of long-distance runners: a randomized crossover clinical trial. Front Nutr. 2025 Aug 13;12:1630462. doi: 10.3389/fnut.2025.1630462. eCollection 2025. PMID 40880737